CLINICAL TRIAL: NCT02793284
Title: Advanced Prostate Imaging of Recurrent Cancer After Radiotherapy
Acronym: PICs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Institute for Cancer Research (Other)
Responsible Party: Principal Investigator, Glenn Bauman, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PICs
Record Dates: First submitted 2016-05-26; First posted 2016-06-08 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention 18F-DCFPyL PET/CT (Experimental): 18F-DCFPyL PET/CT scan obtained at the time of restaging for biochemical recurrence after primary radiotherapy
  Interventions: Radiation: 18F-DCFPyL PET/CT scan

INTERVENTIONS:
Radiation: 18F-DCFPyL PET/CT scan — PET/CT scan using the radioactive agent 18F-DCFPyL

SUMMARY:
The investigators are attempting to determine if a new form of imaging called 18F-DCFPyL PET/CT is helpful to physicians in deciding how to manage suspected prostate cancer recurrence. This imaging uses a Positron Emission Tomography/Computed Tomography (PET/CT) scan using a radioactive tracer 18F-DCFPyL that is concentrated in prostate cancer cells and can potentially identify cancer cells throughout the body. The combination of 18F-DCFPyL PET/CT can potentially identify areas of prostate cancer recurrence not seen with usual imaging [bone scan, computed tomography (CT) thorax, abdomen and pelvis, plus multi-parametric magnetic resonance imaging (MRI)].

DETAILED DESCRIPTION:
The study will evaluate the utility of investigational restaging with 18F-DCFPyL PET/CT following conventional imaging (bone scan, CT thorax, abdomen and pelvis plus multi-parametric pelvic MRI) in detecting the prevalence of metastatic disease among men with biochemical recurrence after radical radiotherapy treatment to the prostate. Men treated with primary radiation with external beam or brachytherapy will be eligible. Eighty (80) eligible consenting patients with biochemical recurrence and potentially suitable for local salvage or targeted ablative therapies will be registered and imaged with conventional imaging (bone scan, CT thorax, abdomen and pelvis plus multi-parametric pelvic MRI) followed by investigational restaging with 18F-DCFPyL PET/CT. Characterizing sites of disease identified by the combination of 18F-DCFPyL PET/CT with conventional imaging versus 18F-DCFPyL PET/CT alone will be used to explore the potential of 18F-DCFPyL PET/CT as a single restaging study in men with biochemical recurrence. While further investigation and treatment after restaging will be at the discretion of the investigator and the patient, the actual treatment/management, treatment outcomes and quality of life will be recorded in an electronic database at 6, 12, 24 and 36 months after re-staging. Such longitudinal analyses of management and outcomes will be useful in characterizing the disease trajectory, response to treatment and quality of life for patients whose recurrent disease is managed based on comprehensive restaging using the combination of conventional imaging and 18F-DCFPyL PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Previous external beam radiotherapy or brachytherapy for localized disease (T1-T2, Gleason < 7 and PSA < 20) or (T1-2, Gleason 8, prostatic specific antigen (PSA)<10)
* Interval to biochemical failure more than 12 months from last radical therapeutic intervention
* Biochemical failure confirmed on at least 3 consecutive PSA measurements each taken at least 1 month apart
* PSA at time of enrollment more than nadir+2.0ng/ml (Phoenix definition of biochemical failure)
* Karnofsky performance status 70 or better [Eastern Cooperative Oncology Group (ECOG) 0,1]
* Total serum testosterone level >1nmol/l (if prior treatment with hormone therapy)

Exclusion Criteria:

* CT or bone scan within 6 months of enrollment
* Patients whose prior radiotherapy was delivered with palliative intent
* Patients with known metastatic disease
* Extensive co-morbidities precluding potential ablative salvage procedures
* Prior history of invasive non-cutaneous malignant disease unless disease free for at least 5 years
* Already on systemic anticancer treatment (androgen deprivation or chemotherapy)
* Inability to comply with the imaging requirements e.g. inability to lie supine for one hour
* Allergy or contraindication to MRI or CT contrast agents or PET tracer to be used as part of the imaging
* Insufficient renal function [estimated glomerular filtration rate (eGFR) < 30 mL/min]

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Detection of extra-prostatic disease | 2 weeks post re-staging
  Number of men with extra-prostatic disease detected by either 18F-DCFPyL PET/CT or conventional imaging, divided by the number of men undergoing imaging.

SECONDARY OUTCOMES:
Detection of extra-prostatic disease exclusive to 18F-DCFPyl PET/CT | 2 weeks post re-staging imaging
  Number of men who have extra-prostatic disease detected exclusively on 18F-DCFPyL PET/CT.
Detection of lesions per subject and overall population | 2 weeks post re-staging imaging
  The number of extra-prostatic lesions detected by 18F-DCFPyL PET/CT versus conventional imaging alone will be compared on a per subject and overall population basis.
Location of extra-prostatic lesions | 2 weeks post re-staging imaging
  The location of extra-prostatic lesions detected by 18F-DCFPyL PET/CT versus conventional imaging.
Planned treatment management based on re-staging imaging | 2 weeks post re-staging imaging
  Planned treatment management based on the information from 18F-DCFPyL PET/CT compared to conventional imaging, to characterize the impact on patient care.
Actual treatment management assessed by physician completed study specific questionnaire | 6 months, 12 months, 24 months, and 36 months after re-staging imaging
  A questionnaire developed specifically for the study, called the Post-PET Management Form, will be completed by the attending physician, noting any changes to the treatment based on the results of the 18F-DCFPyL PET/CT imaging. Treatment options may include, but are not limited to, surgery, radiotherapy, androgen deprivation therapy, cryotherapy, and observation.
Disease status (Is the patient alive, deceased, has active disease, or no evidence of disease?) | 6 months, 12 months, 24 months, and 36 months after re-staging imaging
  The investigators want to determine if the patient is alive, deceased, has active disease or no evidence of disease, at approximately yearly intervals. The source of this data could come from physician notes, lab tests, imaging reports, pathology report, or directly from the patient.
Quality of Life | 6 months, 12 months, 24 months, and 36 months after re-staging imaging
  Quality of life is measured using the Functional Assessment of Cancer Therapy - Prostate (FACT-P) and Expanded Prostate Cancer Index Composite (EPIC) standardized questionnaires.
Disease burden measured by serum and urine biomarkers versus imaging | Baseline
  Baseline serum and urine will be obtained for future correlative studies of novel biomarkers of disease burden for comparison against measures of disease burden provided by imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Bauman, MD, Principal Investigator — London Regional Cancer Program of the Lawson Health Research Institute
Locations (4):
- Canada (4):
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Toronto Sunnybrook Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No